CLINICAL TRIAL: NCT03805425
Title: Photorefractive Intrastromal Corneal Crosslinking (PiXL) for Correction of Hyperopia
Brief Title: PiXL for Correction of Hyperopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gemini Eye Clinic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PiXLHyperopia
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2019-05

CONDITIONS: Hyperopia
Keywords: Hypeorpia; Crosslinking; PiXL
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photorefractive intrastromal corneal crosslinking (PiXL) (Experimental): Patients undergo PiXL where the UVA light is delivered in customized patterns and corneal changes are achieved. For hyperopia, a ring shape irradiation is used to steepen the central cornea. An oxygen mask is used to enhance the crosslinking efficacy. A dedicated riboflavin formulation penetrates the corneal stroma. Pulsed UVA light with oxygen triggers the covalent bonds of collagen strands in riboflavin soaked cornea.
  Interventions: Radiation: PiXL

INTERVENTIONS:
Radiation: PiXL — The system is set to deliver 30 mW/cm2 UVA irradiance in pulsed intervals of 1 second on and 1 second off to 5 to 9 mm diameter corneal annulus. Total energy delivered is 15J.

SUMMARY:
This clinical study aims to investigate the efficacy and safety of PiXL in the refractive correction of low hyperopia.

DETAILED DESCRIPTION:
This clinical study aims to investigate the efficacy and safety of PiXL in the refractive correction of low hyperopia.Slightly modified settings from previously published study is applied to eyes with low hyperopia with an expected refractive change of 0.75 D. Aim is to evaluate the refractive outcome of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* low hyperopia of spherical equivalent from +0.5 up to +1.75 D sp. eq.
* astigmatism up to 0.75 Dcyl
* corneal thickness above 400 µm
* endothelial cell density above 1500 cell/mm2

Exclusion Criteria:

* any prior corneal surgery or any eye surgery within the last 3 months,
* any corneal pathology e.g. corneal scar or dystrophy
* unstable refraction
* patient not able to understand and sign informed consent
* patients with connective tissue disorder or uncontrolled diabetes
* pregnant or lactating women
* aphakic eyes or pseudophakic eyes without UV blocking IOL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in Uncorrected Distance Visual Acuity | Month 12
  Best distance visual acuity tested without any correction
Change in Subjective Refraction | Month 12
  Spherical and cylindrical correction

SECONDARY OUTCOMES:
Change in keratometry | Month 12
  Change in keratomery parameter K2-K1provided by Pentacam
Change in Higher Order Aberrations | Month 12
  Higher Order Aberrations assessed using Pentacam
Change in pachymetry | Month 12
  Change in mean cornea thickness in 8.0 mm ring provided by Pentacam
Subjective questionnaire score | Month 12
  Questionnaire assessing participants discomfort at 6 months in respect to their photophobia, pain and dry eye.
Change in Corrected Distance Visual Acuity | Month 12
  Best distance visual acuity tested with the best correction
Change in Spherical aberration | Month 12
  Spherical aberration assessed using Pentacam

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, MD, PhD, Principal Investigator — Gemini Eye Clinic
Locations (1):
- Gemini Eye Clinic, Zlín, Czechia

REFERENCES:
- [Background] Kanellopoulos AJ, Asimellis G. Hyperopic correction: clinical validation with epithelium-on and epithelium-off protocols, using variable fluence and topographically customized collagen corneal crosslinking. Clin Ophthalmol. 2014 Dec 2;8:2425-33. doi: 10.2147/OPTH.S68222. eCollection 2014. PMID 25506204